CLINICAL TRIAL: NCT00754624
Title: A Four-year, Safety and Tolerability, Open-Label, "Follow on" Trial Evaluating Technosphere® Insulin in Subjects With Type 2 Diabetes Mellitus.
Brief Title: An Open-label, Multi-center, International, Three-year, Safety and Tolerability 'Follow on' Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-010
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (1):
- TI Inhalation Powder (Experimental): Technosphere® Insulin Inhalation Powder
  Interventions: Drug: Technosphere® Insulin Inhalation Powder and MedTone™ Inhaler

INTERVENTIONS:
Drug: Technosphere® Insulin Inhalation Powder and MedTone™ Inhaler — Inhalation starting at 15, 30, or 60U doses and can be titrated up or down by 15U to a minimum of 15U or a maximum of 90U

SUMMARY:
Safety Follow-Up Trial to PDC-INS-0008 and MKC-TI-005

DETAILED DESCRIPTION:
This is an uncontrolled study without comparator. Subjects were followed up to 4 years on Technosphere Insulin. Of 229 subjects 199 were exposed for ≥12 mo, 175 for ≥ 24 mo, 60 for ≥ 36 mo, 31 for ≥ 42 mo, & 2 for 48 mo.

ELIGIBILITY:
Inclusion Criteria:

* Previous completion of PDC-INS-0008 or MKC-TI-005
* Subjects must be able to attend all scheduled visits and, in the opinion of the Investigator, be able to complete this safety trial
* Subjects must be able to understand English or have access to validated primary language trial documents
* Written informed consent

Exclusion Criteria:

* Drug or alcohol dependency
* Smokers (subjects are expected to remain non-smokers throughout their participation in this trial)
* Known hypersensitivity to the trial drug or to drugs of similar chemical structures
* Anemia (hemoglobin level < 11 g/dL for females or < 12 g/dL for males)
* Evidence of moderate or greater ketones in urine
* Women of childbearing potential practicing inadequate birth control. (Adequate birth control is defined as using oral contraceptives, condoms or diaphragms with spermicide, intrauterine devices, Depo-Provera, contraceptive patches or surgical sterilization)
* Women who are pregnant
* Clinically significant adverse events that remain unresolved from the previous trial and/or clinically significant abnormal laboratory values which are determined by the Investigator or the MKC Medical Monitor to be unsafe or confounding to continued participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2004-05; Primary Completion 2008-06 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Boss, MD, Study Director — Mannkind Corporation
Locations (40):
- United States (17):
  - Dorothy L & James E Frank Diabetes Research Institute, San Mateo, California
  - Sansum Medical Research Institute, Santa Barbara, California
  - Alliance Medical Group of Greater Waterbury, Middlebury, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Soundview Research Associates, Norwalk, Connecticut
  - University of Miami School of Medicine, Miami, Florida
  - Oschner Clinic Foundation, New Orleans, Louisiana
  - International Diabetes Center, Minneapolis, Minnesota
  - Diabetes Care & Information Center of New York, Flushing, New York
  - Diabetes Team Associated, New York, New York
  - Endocrine Research - Physician's East PA, Greenville, North Carolina
  - Your Diabetes Endocrine Nutrition Group, Mentor, Ohio
  - Dallas Diabetes & Endocrine Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Diabetes Institute, San Antonio, Texas
  - Diabetes & Glandular Disease Research Assoc PA, San Antonio, Texas
  - Diabetes Care Center, Seattle, Washington
- Bulgaria (8):
  - MBAL "Pleven", Pleven, BGR
  - SBALENG-Sofia Institute of Endocrinology, Sofia, BGR
  - MBAL Alexandrovska Hospital, Sofia, BGR
  - Military Medical Academy, Sofia, BGR
  - Central Clinical Base, Sofia, BGR
  - MBAL "Sweta Marina" - Varna, Varna, BGR
  - II-nd MBAL, Sofia, Sofia
  - Military Medical Academy, Sofia
- Czechia (14):
  - Military Hospital in Brno, Brno, CZE
  - Hospital of "Milosrdnych brain", Brno, CZE
  - University Hospital in Brno, Brno-Bohunice, CZE
  - Surgery of Diabetology, Mělník, CZE
  - University Hospital of 3rd Faculty, Prague, CZE
  - Surgery of Diabetology Petrovice, Prague, CZE
  - Diabetologicka oridnace, Prague, CZE
  - General Hospital in Prague and 1st Faculty of Medicine of, Prague, CZE
  - Institute for Clinical and Exp Medicine, Prague, CZE
  - Surgery of Diabetology Stodulky, Prague, CZE
  - University Hospital Na Bulovce, Prague, CZE
  - Surgery of Diabetology Slany, Slaný, CZE
  - Surgery of Diabetology Zastavka, Zastavka, Brno, CZE
  - Surgery of Diabetology (Brno), Brno
- ikfe Berlin, Berlin, DEU, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled May 31, 2004 Multi-center international trial conducted in USA, Bulgaria, Czech Republic, and Germany. Conducted in medical offices, hospital clinics, and universities.
Pre-assignment Details: This was a follow-on trial for subjects who completed one of the two parent trials (PDC-IND-0008 or MKC-TI-005). Inclusion/Exclusion was participation in these parent trials.
Period: Overall Study
Arm/Group | TI Inhalation Powder
Started | 229
Completed | 160
Not Completed | 69
Not completed — Adverse Event | 16
Not completed — Death | 1
Not completed — Physician Decision | 8
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 28
Not completed — Various | 12
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | TI Inhalation Powder
Number analyzed (Participants) | 229
Age, Continuous [Mean (Full Range); unit: years] | 56.4 [34 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 136
DLCo [Mean (Standard Deviation); unit: mL/min/mmHg] — Lung Diffusion Capacity
  mL/min/mmHg | 26.16 (6.21)
FEV1 [Mean (Standard Deviation); unit: Liters] — Forced Expiratory Volumne in 1 sec.
  Liters | 2.99 (0.70)
FPG [Mean (Standard Deviation); unit: mg/dL] — Fasting Plasma Glucose
  mg/dL | 167.7 (42.1)
FVC [Mean (Standard Deviation); unit: Liters] — Forced Vital Capacity
  Liters | 3.85 (0.89)
HbA1c [Mean (Standard Deviation); unit: %] — Glycosylated Hemoglobin
  % | 7.97 (1.20)
Weight [Mean (Standard Deviation); unit: kg] — Weight in kg
  kg | 87.2 (15.2)

OUTCOME MEASURES:

1. Primary Outcome: Annual Rate of Change in FEV1 From Baseline to End of Study
Time Frame: Baseline to 48 months
Population: Safety Population defined as all subjects who received at least one dose of study drug
Measure: Mean (Standard Error); unit: Liters per year
Arm/Group | TI Inhalation Powder
Number analyzed (Participants) | 229
Liters per year | -0.048 (0.006)
Statistical Analysis 1: Comparison: TI Inhalation Powder; A random coefficient model with a random intercept and slope associated with each subject, was fitted (using the PROC MIXED procedure in SAS) to the observed FEV1 data to estimate the annual rate of decline. The model included terms for baseline FEV1 and time (in years) of FEV1 measurements. Missing pulmonary functions were not imputed; Test type: Superiority or Other; Random coefficient; Adjusted for Baseline FEV1 value; Slope = -0.048, 95% CI 2-sided [-0.059 to -0.037]

2. Secondary Outcome: Annual Rate of Change in FVC From Baseline to End of Study
Time Frame: Baseline to 48 months
Population: Safety
Measure: Mean (Standard Error); unit: Liters per year
Arm/Group | TI Inhalation Powder
Number analyzed (Participants) | 229
Liters per year | -0.058 (0.007)
Statistical Analysis 1: Comparison: TI Inhalation Powder; A random coefficient model with a random intercept and slope associated with each subject, was fitted (using the PROC MIXED procedure in SAS) to the observed FVC data to estimate the annual rate of decline. The model included terms for baseline FVC and time (in years) of FVC measurements. Missing pulmonary functions were not imputed; Test type: Superiority or Other; Random Coefficient; Adjusted for Baseline FVC value; Slope = -0.058, 95% CI 2-sided [-0.072 to -0.043]

3. Secondary Outcome: Annual Rate of Change in DLCo From Baseline to End of Study
Time Frame: Baseline to 48 months
Population: Safety
Measure: Mean (Standard Error); unit: mL/min/mmHg per year
Arm/Group | TI Inhalation Powder
Number analyzed (Participants) | 229
mL/min/mmHg per year | -0.311 (0.073)
Statistical Analysis 1: Comparison: TI Inhalation Powder; A random coefficient model with a random intercept and slope associated with each subject, was fitted (using the PROC MIXED procedure in SAS) to the observed DLco data to estimate the annual rate of decline. The model included terms for baseline DLco and time (in years) of DLco measurements. Missing pulmonary functions were not imputed; Test type: Superiority or Other; Random Coefficient; Adjusted for Baseline DLCo value; Slope = -0.311, 95% CI 2-sided [-0.454 to -0.168]

4. Secondary Outcome: Change in HbA1c From Baseline to Last Measurement on Study Drug (Maximum of 48 Months)
Description: Change in HbA1c from Baseline to last measurement on study drug (maximum of 48 months)
Time Frame: Baseline to last measurement on study drug (maximum of 48 months
Population: Safety
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | TI Inhalation Powder
Number analyzed (Participants) | 225
percentage | 0.20 (1.20)

5. Secondary Outcome: Change in FPG From Baseline to Last Study Measurement on Treatment (Maximum of 48 Months)
Description: Change from Baseline to last study measurement on treatment (maximum of 48 months)
Time Frame: Baseline to last study measurement on treatment (maximum of 48 months)
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | TI Inhalation Powder
Number analyzed (Participants) | 225
milligrams per deciliter | -5.34 (51.43)

6. Secondary Outcome: Change in Weight in kg From Baseline to End of Study
Description: Baseline to last measurement on study drug (maximum of 48 months)
Time Frame: Baseline to last measurement on study drug (maximum of 48 months)
Population: Safety
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | TI Inhalation Powder
Number analyzed (Participants) | 229
kilograms | 1.42 (4.41)

7. Secondary Outcome: High Resolution Computerized Tomography Scans of the Chest
Time Frame: End of study
Population: participants in Safety population with available post-baseline data
Measure: Number; unit: participants
Arm/Group | TI Inhalation Powder
Number analyzed (Participants) | 206
participants
  "Normal" HRCT subjects | 47
  "Abnormal, clinically not significant" subjects | 147
  "Abnormal, Clinically Significant" HRCT subjects | 12

ADVERSE EVENTS:
Time Frame: May 31, 2004 to June 5, 2008
Arm/Group | TI Inhalation Powder
Serious Adverse Events (participants affected / at risk) | 30/229
Other Adverse Events (participants affected / at risk) | 156/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TI Inhalation Powder (N=229)
Anaemia (Blood and lymphatic system disorders) | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 1
Coronary artery disease (Cardiac disorders) | 3
Myocardial ischaemia (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Cardiovascular disorder (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Cataract (Eye disorders) | 1
Appendicitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Device failure (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 1
Localised osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ataxia (Nervous system disorders) | 1
Diabetic neuropathy (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Aortic aneurysm (Vascular disorders) | 1
Arterial stenosis (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TI Inhalation Powder (N=229)
Cataract (Eye disorders) | 12
Diabetic retinopathy (Eye disorders) | 13
Upper respiratory tract infection (Infections and infestations) | 40
Nasopharyngitis (Infections and infestations) | 32
Sinusitis (Infections and infestations) | 13
Bronchitis (Infections and infestations) | 12
Hypoglycaemia (Metabolism and nutrition disorders) | 94
Hypercholesterolaemia (Metabolism and nutrition disorders) | 17
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 19
Back pain (Musculoskeletal and connective tissue disorders) | 18
Headache (Nervous system disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 40
Productive cough (Respiratory, thoracic and mediastinal disorders) | 25
Hypertension (Vascular disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MannKind has right to 1st joint multicenter publication. After 1st publication PI may publish data only if PI submits proposed publication to MNKD for review 60 days prior to publication date. MNKD may remove any confidential information. If a multicenter publication is not submitted 12 months after conclusion, abandonment, or termination of the Study at all sites, or if MNKD confirms there will be no multicenter Study publication, PI may publish the Study results subject to MNKD rights herein.